CLINICAL TRIAL: NCT04291157
Title: Implementability and Health Impact of Proactive Cardiovascular Prevention Strategy in Subjects With High Genetic Risk: a Randomized Pilot Study
Brief Title: Proactive Cardiovascular Prevention Strategy in Subjects With High Genetic Risk
Acronym: EstPerMedCV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Alar Irs (Other)
Collaborators: North Estonia Regional Hospital (Unknown); Tartu University Hospital (Other)
Responsible Party: Sponsor-Investigator, Alar Irs, Teaching physician in cardiology, University of Tartu
Organization: University of Tartu (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EstPerMed CV
Record Dates: First submitted 2020-02-19; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Diseases; Primary Prevention
Keywords: Polygenic risk score
MeSH Terms: conditions — Cardiovascular Diseases; Genetic Risk Score

STUDY DESIGN:
Intervention Model Description: Large simple randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive CVD prevention (Experimental): Proactive invitation to total CVD risk estimation incorporating the PRS and provision of guideline based preventive interventions.
  Interventions: Other: CVD risk estimation incorporating the PRS and guideline based preventive interventions.
- Usual care (Active Comparator): Usual GP care (opportunistic CVD risk estimation and prevention upon usual GP contacts).
  Interventions: Other: Standard GP care

INTERVENTIONS:
Other: CVD risk estimation incorporating the PRS and guideline based preventive interventions. — Total CVD risk estimation using SCORE plus PRS and European Society of Cardiology (ESC) CVD prevention guideline based interventions.
  Arms: Proactive CVD prevention
Other: Standard GP care — Usual GP care (opportunistic CVD prevention)
  Arms: Usual care

SUMMARY:
A polygenic risk score (PRS) will be developed and implemented into the primary care digital work-flow.

1000 study subjects with no known cardiovascular disease, diabetes or statin treatment and with high PRS (men of 30-65, women of 40-70 years of age) will be recruited from amongst the gene donors of Estonian Biobank (Estonian Genome Center at the University of Tartu).

Subjects will be randomised to proactive primary preventive intervention incorporating provision of PRS information or usual care (opportunistic preventive strategy).

Subjects in intervention group will be actively contacted and invited to a general practitioner (GP) based prevention intervention of total cardiovascular risk scoring and guideline recommended preventive measures.

Subjects in control group will be observed for 12 month and then invited to a GP visit and provided the same information and advice as the intervention group.

The impact of PRS on total 10 year cardiovascular disease (CVD) risk scoring will be assessed, the change in total 10 year CVD risk during the intervention will be measured and the difference in total 10 year CVD risk between the groups at month 12 will be reported. Satisfaction of subjects and GPs with the intervention will also be assessed as well as cost-effectiveness of the intervention.

DETAILED DESCRIPTION:
A polygenic risk score (PRS) will be developed and implemented into the primary care digital work-flow.

1000 study subjects with no known cardiovascular disease, diabetes or statin treatment and with high PRS (men of 30-65, women of 40-70 years of age) will be recruited from amongst the gene donors of Estonian Biobank (Estonian Genome Center at the University of Tartu).

Subjects will be randomised to proactive primary preventive intervention incorporating provision of PRS information or usual care (opportunistic preventive strategy).

Subjects in intervention group will be actively contacted and invited to a GP based prevention intervention of total cardiovascular risk scoring and guideline recommended preventive measures.

Subjects in control group will be observed for 12 month and then invited to a GP visit and provided the same information and advice as the intervention group.

The impact of PRS on total 10 year CVD risk scoring will be assessed, the change in total 10 year CVD risk during the intervention will be measured and the difference in total 10 year CVD risk between the groups at month 12 will be reported. Satisfaction of subjects and GPs with the intervention will also be assessed as well as cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male 30-65 years or female 40-70 years
* No history of ischemic heart disease, stroke, TIA or PAD in electronic health record
* No cholesterol lowering treatment
* No history of diabetes
* High PRS of CVD
* No physical or mental conditions precluding informed consent or participation

Exclusion Criteria:

* History of ischemic heart disease, stroke, transitory ischemic attack (TIA) or peripheral artery disease (PAD) in electronic health record
* Cholesterol lowering treatment
* History of diabetes
* No consent to participate

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Total 10 year cardiovascular disease (CVD) risk | 12 months
  SCORE (Systematic COronary Risk Evaluation), estimates fatal cardiovascular disease events over a ten-year period in %.
  Employs categories of 1) low (calculated SCORE <1%) 2) moderate-risk (calculated SCORE1% to <5%), 39 ) high-risk (calculated SCORE5% to <10%) and 3) very-high-risk (calculated SCORE ≥10%).
  Conroy RM , Pyorala K, Fitzgerald AP et al. Estimation of ten-year risk of fatal cardiovascular disease in Europe: the SCORE project. Eur H J2003;24:987-1003.

SECONDARY OUTCOMES:
Treatment initiation (first prescription) or dose escalation (new prescription with a higher dose) of CVD preventive pharmacotherapy | 12 months
  New prescription or a dose escalation of any anti-hypertensive, lipid lowering, anti-platelet or anti-smoking medicinal product.
Adherence to CVD prevention recommendations | 12 months
  Adherence to CVD prevention recommendations - proportion of patients adhering to lifestyle advice as recorded by GP.
Systolic blood pressure | 12 months
  Sitting systolic blood pressure measured by automated device at GP office, mmHg
Diastolic blood pressure | 12 months
  Sitting diastolic blood pressure measured by automated device at GP office, mmHg
Total cholesterol | 12 months
  mmol/L
LDL cholesterol | 12 months
  mmol/L
BMI | 12 months
  Body mass index, height (m) and weight (kg) combined (kg/m2)
Waist circumference | 12 months
  cm, measured at GP office
Smoking status | 12 months
  Self-reported smoking status as recorded at GP office
Physical activity | 12 months
  Self-reported physical activity, min/week, as recorded at GP office
Satisfaction of gene donors with intervention | 12 months
  Satisfaction of gene donors with intervention - descriptive questionnaire, analysed qualitatively
Satisfaction of GPs with intervention | 12 months
  Satisfaction of GPs with intervention - descriptive questionnaire, analysed qualitatively
Cost-effectiveness of intervention | 12 months, modelled over lifetime
  Incremental cost-effectiveness ratio (EUR/QALY): cost of intervention combined in an economic model with lifetime benefit (number of quality adjusted life years modelled based on change in total CVD risk, measured as primary endpoint).

CONTACTS AND LOCATIONS:
Overall Officials: Margus Viigimaa, MD, PhD, Principal Investigator — University of Tartu
Locations (2):
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Hospital, Tartu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study general information and contacts — https://sisu.ut.ee/pmkliinilisedjuhtprojektid